CLINICAL TRIAL: NCT02612415
Title: FIRST-ABC Feasibility Study: Feasibility Study for a Randomised Trial of High Flow Nasal Cannula (HFNC) Versus Continuous Positive Airway Pressure (CPAP) for Non-invasive Respiratory Support in Critically Ill Children
Brief Title: FIRST-line Support for Assistance in Breathing in Children (FIRST-ABC) Feasibility Study
Acronym: FIRST-ABC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); Barts & The London NHS Trust (Other); Intensive Care National Audit & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14HC30
Record Dates: First submitted 2015-10-23; First posted 2015-11-23 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Hypoxia; Respiratory Acidosis; Moderate/Severe Respiratory Distress
MeSH Terms: conditions — Hypoxia; Acidosis, Respiratory; Lymphoma, Follicular; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flow nasal cannula (HFNC) (Experimental): Heated humidified high flow nasal cannula therapy delivered at 2 L/kg/min gas flow rate (for children older than 10 kg in weight, an additional 0.5 L/kg/min per kilogram over 10 kg). Any approved device can be used to deliver HFNC
  Interventions: Device: Treatment strategy: Non-invasive respiratory support delivered via high flow nasal cannula
- Continuous positive airway pressure (CPAP) (Active Comparator): Continuous positive airway pressure delivered using any interface (hood, mask or prongs)
  Interventions: Device: Treatment strategy: Non-invasive respiratory support delivered via continuous positive airway pressure

INTERVENTIONS:
Device: Treatment strategy: Non-invasive respiratory support delivered via high flow nasal cannula — A heated, humidified, HFNC device will be used to deliver a gas flow rate of 2 L/kg/min for the duration that the patient needs non-invasive respiratory support
  Arms: High flow nasal cannula (HFNC)
Device: Treatment strategy: Non-invasive respiratory support delivered via continuous positive airway pressure — CPAP will be provided using a set expiratory pressure of 6-8 cm water (H2O) pressure for the duration that the infant needs non-invasive respiratory support
  Arms: Continuous positive airway pressure (CPAP)

SUMMARY:
A feasibility study to inform the design and conduct of a randomised controlled trial of high flow nasal cannula (HFNC) versus continuous positive airway pressure (CPAP) for non-invasive respiratory support in critically ill children

DETAILED DESCRIPTION:
Breathing support is the most common intervention provided to critically ill children in a paediatric intensive care unit (PICU). Although invasive breathing support (delivered through a tracheal tube) is lifesaving, concerns regarding its risks (infection and lung damage) have prompted greater use of non-invasive respiratory support (NRS). However, there is little scientific evidence to guide PICU clinicians on the comparative effectiveness of the commonly used modes of NRS.

In this feasibility study, the investigators are testing whether it is possible to conduct a randomised clinical trial comparing two modes of NRS: continuous positive airway pressure (CPAP), which has been used for over two decades, and high flow nasal cannula (HFNC), a newer method of respiratory support. It is not known for sure how useful HFNC is in critically ill children because there is no published research comparing it with CPAP. However, since HFNC is easier to use and better tolerated by children, many hospitals are now using HFNC instead of CPAP. Before HFNC is widely adopted, a clinical trial to establish its role in the management of critically ill children is urgently needed.

As part of this study, the investigators will randomly allocate children deemed to require NRS by their treating clinician to either HFNC or CPAP. The investigators will mainly assess whether sufficient number of children can be recruited to the trial, whether clinicians are willing to randomise children, and test the proposed treatment pathways for CPAP and HFNC. The trial will run over six months, and recruit 120 sick children from three National Health Service (NHS) hospitals. Consent will be sought from parents/guardians for their children to be included in the study, usually before CPAP or HFNC is started, unless emergency life-saving treatment is required, in which case consent will be deferred until there is more time to discuss the study with parents/guardians.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will fall into one of two groups:

Group A (Step-up)

1. Age >36 weeks corrected gestational age and <16 years, AND
2. Deemed to require non-invasive respiratory support by the treating clinician for an acute illness, AND
3. Satisfies one or more of the following criteria:

   * Hypoxia (oxygen saturation <92% in fraction of inspired oxygen (FiO2) >0.40, or equivalent). FiO2 of 0.40 roughly equates to standard unhumidified nasal cannula oxygen delivered at 6 L/min or oxygen delivered via facemask without a rebreather bag at 6-10 L/min.
   * Acute respiratory acidosis (pH <7.3 with a concomitant pCO2 >6.5 kPa)
   * Moderate respiratory distress (use of accessory muscles, subcostal and intercostal recession, tachypnoea for age, grunting)

Group B (Step-down)

1. Age >36 weeks corrected for gestation and <16 years, AND
2. Deemed to require non-invasive respiratory support by the treating clinician after extubation, following a spell of invasive ventilation

   * Either immediately after extubation as a 'planned' procedure, irrespective of clinical condition ('planned') OR
   * Prompted by deterioration in clinical condition within 72 hours after extubation ('rescue'). Clinical parameters to assess the need for NRS in this situation will be similar to point 3 in Group A.

Exclusion Criteria:

1. Deemed by the treating clinician to require immediate intubation/invasive ventilation due to severe hypoxia, acidosis and/or respiratory distress, upper airway obstruction or recurrent apnoeas
2. Tracheostomy in place
3. Pre-existing air-leak syndrome (pneumothorax/pneumomediastinum)
4. Midfacial/craniofacial anomalies (unrepaired cleft palate, choanal atresia) or had recent craniofacial surgery
5. Agreed limitation of intensive care treatment plan in place ('not for intubation')
6. On domiciliary non-invasive ventilation prior to PICU admission
7. Managed on either HFNC and/or CPAP (or other form of non-invasive ventilation such as BiPAP) in the preceding 24 hours
8. Previously recruited to this study during the same PICU admission
9. Cannot be treated with HFNC

   * Unavailability of appropriate sized nasal prongs
   * Unavailability of HFNC device
10. Cannot be treated with CPAP

    * Unavailability of right size of face mask, prong or other patient interface
    * Unavailability of CPAP device

Ages: 36 Weeks to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients in Group A (step-up) and Group B (step-down) | Baseline
Number of parents/guardians who refuse prospective or deferred consent | Through study completion, an average of 24 hours
Randomising at least 50% of eligible patients | Baseline
Proportion of patients adherent to the study treatment | Through study completion, an average of 72 hours
Mean COMFORT score | 72 hours
Number of parents completing the Parental Stressor Scale: PICU (PSS:PPICU) | 24 hours

SECONDARY OUTCOMES:
Proportion of children randomised to the intervention or control who need intubation (Group A) or re-intubation (Group B) | 72 hours
Proportion of children randomised to the intervention or control who fail the assigned treatment and require either crossover or escalation to other forms of ventilation | 72 hours
Number of children who experience pre-specified adverse events (pneumothorax, pneumomediastinum, nasal or facial trauma, abdominal distension, nosocomial infection) during the period they are receiving non-invasive respiratory support | 28 days
Improvement in oxygenation, partial pressure of carbon dioxide (pCO2) levels, heart rate, respiratory rate, and work of breathing | 24 hours
Length of PICU and hospital stay, length of invasive ventilation, length of non-invasive support, ventilator-free days at day 28 | through study completion, an average of 28 days
Mortality at PICU discharge and at hospital discharge | through study completion, an average of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Padmanabhan Ramnarayan, Principal Investigator — Consultant in Paediatric Intensive Care & Retrieval Children's Acute Transport Service (CATS)
Locations (3):
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Ramnarayan P, Lister P, Dominguez T, Habibi P, Edmonds N, Canter RR, Wulff J, Harrison DA, Mouncey PM, Peters MJ; United Kingdom Paediatric Intensive Care Society Study Group (PICS-SG). FIRST-line support for Assistance in Breathing in Children (FIRST-ABC): a multicentre pilot randomised controlled trial of high-flow nasal cannula therapy versus continuous positive airway pressure in paediatric critical care. Crit Care. 2018 Jun 4;22(1):144. doi: 10.1186/s13054-018-2080-3. PMID 29866165
- [Derived] Ramnarayan P, Lister P, Dominguez T, Habibi P, Edmonds N, Canter R, Mouncey P, Peters MJ. FIRST-line support for Assistance in Breathing in Children (FIRST-ABC): protocol for a multicentre randomised feasibility trial of non-invasive respiratory support in critically ill children. BMJ Open. 2017 Jun 12;7(6):e016181. doi: 10.1136/bmjopen-2017-016181. PMID 28606907